CLINICAL TRIAL: NCT07391878
Title: Open-Label Study to Evaluate the Safety and Efficacy of Two Doses of TRG-200 KIT in Patients With Refractory Overactive Bladder (OAB) : A Pilot Study
Brief Title: Evaluate the Safety and Efficacy of TRG-200 KIT in Patients With Refractory Overactive Bladder.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Trigone Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRGC-05
Record Dates: First submitted 2025-12-22; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Overactive Bladder (OAB)
Keywords: Refractory Overactive Bladder (OAB)
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: Open-label, parallel-assignment study with two experimental dose-evaluation arms (150 mg and 300 mg). An adaptive two-stage design is used for dose selection, followed by expansion with the selected dose.
Who Masked: Participant
Masking Description: This study is primarily open-label. A short single-blind placebo run-in period is conducted prior to treatment initiation, during which participants are blinded to the placebo instillation. Investigators are aware of the treatment administered. All subsequent treatment phases are open-label, with no masking applied.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TRG-200 KIT - 150 mg (Dose-Evaluation Cohort) (Experimental): Participants receive intravesical administration of TRG-200 KIT containing oxybutynin 150 mg. The investigational product is administered via intravesical instillation following a single-blind placebo run-in period. This arm is part of the initial dose-evaluation stage to assess safety, tolerability, and preliminary efficacy.
  Interventions: Drug: TRG-200 KIT
- TRG-200 KIT - 300 mg (Dose-Evaluation Cohort) (Experimental): Participants receive intravesical administration of TRG-200 KIT containing oxybutynin 300 mg. The investigational product is administered via intravesical instillation following a single-blind placebo run-in period. This arm is part of the initial dose-evaluation stage to assess safety, tolerability, and preliminary efficacy.
  Interventions: Drug: TRG-200 KIT

INTERVENTIONS:
Drug: TRG-200 KIT — TRG-200 KIT is administered intravesically as a sustained-release formulation. The investigational product consists of a Carbopol gel matrix followed by intravesical instillation of oxybutynin via a urethral catheter, forming a prolonged-release delivery system within the bladder.
  The intervention is designed to provide sustained local bladder exposure while minimizing systemic absorption and anticholinergic adverse effects.

SUMMARY:
This is an open-label, single-center pilot study designed to evaluate the safety, tolerability, and preliminary efficacy of TRG-200 KIT, an intravesical sustained-release oxybutynin formulation, in adult patients with refractory overactive bladder (OAB). The study includes an adaptive two-stage design with initial dose evaluation of two dose levels (150 mg and 300 mg oxybutynin) followed by expansion using the selected dose. TRG-200 KIT is administered via monthly intravesical instillation and aims to provide prolonged local bladder exposure while minimizing systemic absorption and anticholinergic adverse effects.

DETAILED DESCRIPTION:
Overactive bladder (OAB) is a prevalent chronic condition characterized by urinary urgency, usually accompanied by increased frequency and nocturia, with or without urgency urinary incontinence. Despite the availability of behavioral, pharmacologic, and invasive therapies, a substantial proportion of patients remain refractory or intolerant to current treatments, particularly oral antimuscarinic agents due to systemic side effects and limited long-term adherence.

This open-label, pilot clinical study (TRGC-05) is designed to evaluate the safety, tolerability, efficacy, and exploratory pharmacokinetics of TRG-200 KIT, a novel intravesical sustained-release delivery system containing oxybutynin. TRG-200 KIT consists of a Carbopol gel matrix followed by intravesical administration of oxybutynin (150 mg or 300 mg), forming a prolonged-release system within the bladder to enhance local therapeutic exposure while reducing systemic absorption.

The study employs an adaptive two-stage design. In Stage 1, approximately 20 participants are enrolled into two sequential dose-evaluation cohorts (10 participants per dose level: 150 mg and 300 mg). Safety, tolerability, and pharmacokinetic data from these participants are reviewed to select the optimal dose. In Stage 2, approximately 30 additional participants are treated with the selected dose to further characterize safety and efficacy.

All participants undergo screening, a single-blind placebo run-in period, and an open-label treatment phase consisting of three monthly intravesical instillations of TRG-200 KIT, followed by post-dose endpoint and end-of-study assessments. Efficacy is primarily evaluated by changes from baseline in micturition frequency and other OAB symptoms using patient voiding diaries and validated questionnaires, including quality-of-life measures. Safety assessments include adverse event monitoring, laboratory tests, vital signs, physical and urological examinations, and post-void residual volume measurements. Exploratory pharmacokinetic assessments are performed in a subset of participants to characterize systemic exposure to oxybutynin following intravesical administration.

The study is conducted at Shaare Zedek Medical Center in Jerusalem, Israel, and is intended to inform dose selection and support further clinical development of TRG-200 KIT as a potential treatment option for patients with refractory OAB.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent and comply with all study procedures.
2. Male or female adults aged 18 years or older.
3. Documented diagnosis of overactive bladder (OAB) for more than 6 months, refractory or intolerant to oral anticholinergic or other OAB therapies.

   OAB is defined as urinary urgency, usually accompanied by frequency and/or nocturia, with or without urgency urinary incontinence.
4. Ability to perform and tolerate urethral catheterization for intravesical instillation.
5. Meets the following criteria based on the 3-day voiding diary completed at both the Run-in and Baseline visits:

   1. Average of ≥8 micturitions per day, and
   2. Average of ≥3 urgency episodes per day, and
   3. Average of ≥2 nocturia episodes per night.
6. Participants who report significant improvement during the Run-in phase may continue in the study, provided they meet all inclusion criteria, following consultation with the investigator and based on their self-reported assessment.
7. Post-void residual (PVR) urine volume <150 mL.
8. Negative urine culture at screening.
9. Women of childbearing potential must have a negative serum pregnancy test at screening and agree to use effective contraception throughout the study.
10. Stable medical condition, without acute illness, as determined by the investigator.
11. Demonstrated ability to complete the 3-day voiding diary as reviewed at the Run-in and Baseline visits.

Exclusion Criteria:

1. Pregnant or breastfeeding women, or women of childbearing potential not using acceptable contraception.
2. Known contraindication, hypersensitivity, or allergy to oxybutynin or other anticholinergic agents.
3. History of 24-hour urine volume >3,000 mL.
4. Active urinary tract infection or genitourinary infection at screening (re-screening allowed once after treatment).
5. Lower urinary tract pathology that may account for symptoms, including but not limited to:

   urethral diverticulum, radiation cystitis, tuberculosis cystitis, neurogenic bladder, vaginal candidiasis, urolithiasis, interstitial cystitis, urothelial tumor, clinically significant benign prostatic hyperplasia with obstruction, bladder outlet obstruction, prostatitis, prostate or gastrointestinal cancer.
6. Structural abnormalities of the bladder (e.g., diverticula, stones) or urogenital anatomical defects.
7. History of bladder tumors or prostate cancer within the past 5 years, or history of non-muscle invasive bladder cancer (low-grade) within the past 5 years.
8. Ongoing or planned treatment for urologic or gynecologic malignancy.
9. Requirement for indwelling catheter or clean intermittent catheterization (CIC), implanted nerve stimulator, or prior procedures affecting bladder function.
10. Renal insufficiency or serum creatinine >1.5 times the upper limit of normal, or patients on dialysis.
11. Recent pelvic surgery or pelvic radiation within the past 6 months.
12. Neurological conditions affecting bladder function or contraindicating catheterization.
13. Alcohol or drug abuse.
14. Uncontrolled diabetes mellitus.
15. Hemodynamic instability, including abnormal heart rate, respiratory rate, blood pressure, or oxygen saturation outside protocol-defined ranges.
16. Unstable cardiovascular disorders, including but not limited to myocardial infarction, ischemic heart disease, atrial fibrillation, heart block, Wolff-Parkinson-White syndrome, bradycardia, coronary artery disease, or QT prolongation.
17. History of significant liver dysfunction, gastrointestinal bleeding, renal disease, seizures, inflammatory bowel disease, or hepatitis.
18. Clinically significant hematologic abnormalities, including leukopenia, thrombocytopenia, or anemia below protocol-defined thresholds.
19. Body mass index (BMI) ≥40 kg/m².
20. Any medical condition that, in the investigator's opinion, may place the participant at increased risk, confound study results, or interfere with study conduct.
21. Recent changes (within 8 weeks) in lower urinary tract interventions, including neuromodulation, tibial nerve stimulation, pelvic floor muscle training, or biofeedback.
22. Lifetime history of psychotic or bipolar disorder.
23. Active genital herpes or vaginitis.
24. Women with urinary symptoms occurring exclusively during menstruation.
25. Participation in another interventional clinical trial within 30 days prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-12-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Average Number of Micturitions per 24 Hours | Baseline to Week 12
  Change from baseline in the average number of micturitions per 24 hours, as recorded in a 3-day patient voiding diary.
Change From Baseline in Average Number of Urgency Episodes per 24 Hours | Baseline to Week 12
  Change from baseline in the average number of urgency episodes (defined as a sudden and compelling desire to void) per 24 hours, based on the 3-day patient voiding diary.
Change From Baseline in Average Number of Urgency Urinary Incontinence (UUI) Episodes per 24 Hours | Baseline to Week 12
  Change from baseline in the average number of urgency urinary incontinence (UUI) episodes per 24 hours, as recorded in the 3-day patient voiding diary.

SECONDARY OUTCOMES:
Proportion of Participants With ≥50% Reduction in Micturitions per 24 Hours | Baseline to Week 12
  Proportion of participants achieving at least a 50% reduction from baseline in the average number of micturitions per 24 hours, based on the 3-day patient voiding diary.
Proportion of Participants With ≥50% Reduction in Urgency Episodes per 24 Hours | Baseline to Week 12
  Proportion of participants achieving at least a 50% reduction from baseline in the average number of urgency episodes per 24 hours, based on the 3-day patient voiding diary.
Proportion of Participants With ≥50% Reduction in Urgency Urinary Incontinence (UUI) Episodes | Baseline to Week 12
  Proportion of participants achieving at least a 50% reduction from baseline in the average number of urgency urinary incontinence (UUI) episodes per 24 hours.
Change From Baseline in Nocturnal Voids per Night | Baseline to Week 12
  Change from baseline in the average number of nocturnal voids per night, as recorded in the 3-day patient voiding diary.
Change From Baseline in Average Voided Volume | Baseline to Week 12
  Change from baseline in average voided volume (mL), measured using a calibrated measuring device and recorded in the patient voiding diary.
Change From Baseline in Quality of Life Score | Baseline to Week 12
  Change from baseline to Week 12 in quality of life related to lower urinary tract symptoms, assessed using the LUTN questionnaire total score.
  The LUTN questionnaire total score ranges from 0 to 100, with higher scores indicating greater symptom burden and poorer quality of life, and lower scores indicating improvement. The outcome measure will be reported as the mean change from baseline.
Improvement in Patient Perception of Bladder Condition (PPBC) | Baseline to Week 12
  Proportion of participants achieving an improvement of at least 1 point on the 6-point Patient Perception of Bladder Condition (PPBC) scale.
Incidence and Severity of Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | From first dose through End of Study (Week 12)
  Incidence, severity, and relationship to study treatment of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) will be assessed from first dose through Week 12. Events will be coded using MedDRA and summarized by system organ class, preferred term, severity (mild, moderate, severe), and relationship to study treatment.
Change From Baseline in Vital Signs (Blood Pressure, Heart Rate, and Body Temperature) | Baseline to Week 12
  Change from baseline to Week 12 in systolic blood pressure (mmHg), diastolic blood pressure (mmHg), heart rate (beats per minute), and body temperature (°C). Results will be summarized as mean change from baseline for each parameter.
Change From Baseline in Clinical Laboratory Safety Parameters | Baseline to Week 12
  Change from baseline to Week 12 in clinical laboratory parameters including hematology (hemoglobin, white blood cell count, platelet count) and serum chemistry (creatinine, ALT, AST). Results will be summarized as mean change from baseline and incidence of values outside the normal reference range.
Change From Baseline in Post-Void Residual Urine Volume | Baseline to Week 12
  Change from baseline to Week 12 in post-void residual (PVR) urine volume, measured in milliliters (mL) using bladder ultrasound. Results will be summarized as mean change from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel